CLINICAL TRIAL: NCT02811822
Title: A Phase I Open-Label Dose Escalation Study to Determine the Efficacy, Safety and Pharmacokinetics of GMI-1271 as Adjunct to Standard of Care Chemotherapy for the Treatment of Multiple Myeloma
Brief Title: A Study to Determine the Efficacy, Safety and Pharmacokinetics of GMI-1271 as Adjunct to Standard of Care for the Treatment of Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlycoMimetics Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GMI-1271-230
Record Dates: First submitted 2016-06-20; First posted 2016-06-23 (Estimated); Last update posted 2019-07-10 (Actual); Status verified 2019-07

CONDITIONS: Multiple Myeloma
Keywords: GMI-1271; bortezomib; carfilzomib; multiple myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — uproleselan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Dose 1 (Experimental)
  Interventions: Drug: GMI-1271
- Dose 2 (Experimental)
  Interventions: Drug: GMI-1271
- Dose 3 (Experimental)
  Interventions: Drug: GMI-1271
- Dose 4 (Experimental)
  Interventions: Drug: GMI-1271

INTERVENTIONS:
Drug: GMI-1271

SUMMARY:
This study will evaluate GMI-1271, a specific E-selectin antagonist, in multiple myeloma as adjunct to standard of care chemotherapy used to treat this disease.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females ≥ 18 years of age
2. Confirmed diagnosis of Multiple Myeloma
3. Subjects with progressive MM who have received at least 1 prior therapy and who have already undergone or are not expected to undergo hematopoietic stem cell transplantation
4. Subjects previously treated with an IMiD-based regimen or ineligible for an IMiD-based treatment regimen
5. Subjects must be receiving treatment with a proteasome inhibitor-based regimen (bortezomib-based or carfilzomib-based)
6. Adequate hepatic, renal, and cardiac function

Exclusion Criteria:

1. Intolerant to bortezomib or carfilzomib
2. Progressing evidence of end organ damage attributed to the underlying disease
3. Plasma cell leukemia
4. Congestive heart failure
5. Acute active infection
6. Non-hematologic malignancy within the past 3 years except: a) adequately treated basal cell or squamous cell skin cancer, b) carcinoma in situ of the cervix, or c) prostate cancer with stable PSA
7. Significant peripheral neuropathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2019-04 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
Safety assessed by frequency, severity and relatedness of AEs | up to 6 months
  Assessed by frequency, severity and relatedness of AEs
Overall Response Rate | up to 18 months
  Overall Response Rate = Stringent Complete Response + Complete Response + Very Good Partial Response + Partial Response

SECONDARY OUTCOMES:
Clinical benefit rate = Stringent Complete Response + Complete Response + Very Good Partial Response + Partial Response + Minimal Response + Stable Disease | 18 months
Time to response | 18 months
Time to progression | 18 months
Duration of response | 18 months
Progression free survival | 18 months
Overall survival | 18 months
Time versus plasma concentration profile of GMI-1271 | up to Day 23 of Cycle 1 (each cycle is 21 or 28 days)

CONTACTS AND LOCATIONS:
Overall Officials: Michael O'Dwyer, MD, Principal Investigator — National University Ireland - Galway
Locations (8):
- Vejle Hospital, Vejle, Denmark
- Medizinische Klinik/Abt. Innere Medizin V, Heidelberg, Germany
- Ireland (3):
  - Cork University Hospital, Wilton, Cork
  - Beaumont Hospital, Dublin
  - National University Ireland - Galway, Galway
- United Kingdom (3):
  - Sheffield Teaching Hospital, Sheffield, England
  - Saint James's University Hospital Leeds, Leeds
  - University College London Hospitals, London

IPD SHARING:
Plan to Share IPD: No